CLINICAL TRIAL: NCT05776134
Title: Expanded Access Study for the Treatment of Patients With Commercially Out-of-Specification Brexucabtagene Autoleucel
Status: Available | Type: Expanded Access
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Other Study IDs: KT-US-472-0141
Record Dates: First submitted 2023-03-03; First posted 2023-03-20 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Mantle Cell Lymphoma; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — brexucabtagene autoleucel

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Brexucabtagene Autoleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells/kg administered intravenously.
  Other Names: Tecartus™

SUMMARY:
The goal of this study is to provide access to brexucabtagene autoleucel for patients diagnosed with a disease approved for treatment with brexucabtagene autoleucel, that is otherwise out of specification for commercial release.

ELIGIBILITY:
Inclusion Criteria:

* Have commercially manufactured brexucabtagene autoleucel that does not meet commercial release criteria but does meet Kite clinical trial release criteria
* Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been post-menopausal for at least 2 years are not considered to be of childbearing potential)
* Deemed medically fit and stable to receive the product per the investigator's evaluation
* Repeat leukapheresis is not feasible per the investigator's assessment
* Be diagnosed with 1 of the approved labeled indications for brexucabtagene autoleucel that is intended for release
* In the Investigator's opinion, there is no satisfactory alternative therapy available to the individual

Exclusion Criteria:

* History of severe immediate hypersensitivity to any drugs or metabolites of similar chemical classes as brexucabtagene autoleucel
* Uncontrolled active infection or inflammation per physician assessment
* Primary central nervous system (CNS) lymphoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (44):
- United States (44):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - St. Luke's Cancer Institute, Boise, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Kansas Medical Center, Westwood, Kansas
  - University of Maryland Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute - Chestnut Hill, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine- Siteman Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medicine - NewYork-Presbyterian Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center (MMC), The Bronx, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sarah Canon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt-Ingrim Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Methodist Healthcare System of San Antonio dba Methodist Hospital, San Antonio, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KT-US-472-0141